CLINICAL TRIAL: NCT05033405
Title: The Effect of Neuro Linguistic Programming on Pain Levels After Cesarean Delivery: A Randomized Controlled Trial
Brief Title: Neuro Linguistic Programming Pain Levels After Cesarean Delivery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Munzur University (Other)
Responsible Party: Principal Investigator, Nursel Alp Dal, Asis. Prof., Munzur University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Supportive Care
Other Study IDs: 047213793060212
Record Dates: First submitted 2021-08-18; First posted 2021-09-02 (Actual); Last update posted 2021-09-02 (Actual); Status verified 2021-08

CONDITIONS: Nursing Caries; Pain, Postoperative
Keywords: NLP, cesarean section, postpartum, pain
MeSH Terms: conditions — Pain, Postoperative; Pain | interventions — Neurolinguistic Programming

STUDY DESIGN:
Intervention Model Description: The study was conducted by using a prospective randomized single-blind clinical trial model.
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental:Neuro Linguistic Programming (Experimental): One session (20-minute long) of NLP application was performed. The NLP techniques that were employed were representational systems and submodality. In this technique, the sensory, auditory, and kinesthetic feelings of the individual are learned. These emotions are modified by imagining. The NLP application was carried out by a researcher who has a certificate in this field.
  Interventions: Behavioral: NEURO-LINGUISTIC PROGRAMMING (NLP)
- control group (No Intervention): No NLP was applied on the control group patients.

INTERVENTIONS:
Behavioral: NEURO-LINGUISTIC PROGRAMMING (NLP) — ● One session (20-minute long) of NLP application was performed. The NLP techniques that were employed were representational systems and submodality. In this technique, the sensory, auditory, and kinesthetic feelings of the individual are learned. These emotions are modified by imagining. The NLP application was carried out by a researcher who has a certificate in this field
  Arms: Experimental:Neuro Linguistic Programming

SUMMARY:
This study was conducted to determine the effect of Neuro-Linguistic Programming (NLP) application on post-cesarean section pain levels.

DETAILED DESCRIPTION:
The study was carried out between March 1 and June 1, 2021 with mothers who gave birth through cesarean section in the postpartum service of a maternity and children's hospital in the most populated city of Turkey, which is located in the west. The study data consists of a total of 76 individuals, including 38 in the experimental group and 38 in the control group. In the study, the effect size was calculated as 2.22. Accordingly, the power of the study, which was completed with 38 individuals in the control group and 38 in experimental group, had an effect size of 2.22, and used a significance level of 0.05, was calculated as 99.9%. The power analysis was conducted on the G*Power software package.

ELIGIBILITY:
Inclusion Criteria:

* The study included individuals who

  * had a cesarean section,
  * were at the 6th to 24th hour postpartum,
  * agreed to participate in the study,
  * had a cesarean section for the first time,
  * did not use patient-controlled analgesia (PCA),
  * did not have an additional health problem that may cause pain in the postpartum period, other than cesarean incision pain, and
  * could speak and understand Turkish.

Exclusion Criteria:

* Mothers who wanted to quit on their own will at any stage after being included in the study, had verbal communication problems, had hearing or vision problems, or had previously been diagnosed with a psychiatric illness were excluded from the sample.

Ages: 19 Years to 42 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — The mothers who gave birth through cesarean section in the postpartum service of a maternity and children's hospital
Enrollment: 76 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2021-06-01 (Actual); Study Completion 2021-06-21 (Actual)

PRIMARY OUTCOMES:
Examination of inter-and intra-group differences regarding VAS Scores | Immediately after the completion of the NLP application
  A mean total score on the Visual Analogue Scale (VAS). In this assessment, users score their pain from 0 to 10. The scores are interpreted as follows: "0", no pain at all; 1-4, mild pain; 5-6, moderate pain; and 7-10, severe pain.
  A mean total score on the VAS of four and above indicates postoperative pain.

SECONDARY OUTCOMES:
Distribution of participant characteristics by groups | 20 minutes after the first administration of the VAS
  The effect of NLP application on post-operative pain in women who gave birth by cesarean section is examined. Comparisons are made by using Visual Analog Scale (VAS) mean scores in the experimental and control groups.

CONTACTS AND LOCATIONS:
Locations (1):
- Nursel Alp Dal, Tunceli, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided